CLINICAL TRIAL: NCT01487993
Title: An Efficacy, Safety and Pharmacokinetic Study on the Short-term and Long-term Use of Metformin in Obese Children and Adolescents
Brief Title: Metformin in Obese Children and Adolescents
Acronym: MetVoorMin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, Van der Vorst, Mrs. M.M.J. van der Vorst, paediatrician-clinical pharmacologist, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Metformin 2011-6; 2010-023980-17 (EudraCT Number)
Record Dates: First submitted 2011-10-20; First posted 2011-12-08 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Insulin Resistance
Keywords: Obesity; Children; Adolescents; Metformin; Insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Metformin with lifestyle intervention during 18 months
  Interventions: Drug: Metformin; Behavioral: Lifestyle intervention
- Placebo (Placebo Comparator): Placebo and lifestyle intervention during 18 months
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Drug: Metformin — Oral administration, 500 mg daily at week 1. Every week metformin dosage increases with 500 mg, to a maximum dose of 1000 mg bid. This maximum dose will be administered till the end of the study.
  Other Names: Glucophage
  Arms: Metformin
Behavioral: Lifestyle intervention — Lifestyle intervention: 18 months physical therapy and dietary advice

SUMMARY:
The purpose of this study is to determine whether metformin is effective in reducing BMI and insulin resistance in obese children and adolescents.

DETAILED DESCRIPTION:
The prevalence of obesity in children and adolescents is increasing rapidly and is associated with significant medical and psychosocial consequences persisting into adulthood.

Obesity may lead to metabolic complications, such as insulin resistance, which can progress via impaired fasted glucose and impaired glucose tolerance to type 2 diabetes mellitus (T2DM) and to the development of micro- and macro-vascular complications.

Metformin, an oral anti-diabetic licensed for T2DM for adults and children from 10 years onwards, is already used off label in obese children and adolescents with insulin resistance, even though the specific effects of metformin in these obese children and adolescents have not been elucidated, particularly upon long-term use.

The rationale for this study is based on the hypothesis that metformin may reduce body mass index (BMI), insulin resistance and percentage of body-fat in obese children and adolescents with insulin resistance. Further more it is anticipated that metformin may delay the progression to T2DM and thereby micro- and macro-vascular complications in obese children and adolescents with insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 10 and ≤ 16 years at study entry
* Caucasian descent
* Obesity defined as BMI-SDS > 2.3
* Insulin resistance defined as HOMA-IR ≥ 3.4.
* An obtained informed consent from subjects and parents/caregivers.

Exclusion Criteria:

* Presence of T2DM (American Diabetes Association criteria)
* Presence of endocrine disorders with steroid therapy
* Suspicion of polycystic ovarium syndrome;
* Height < -1.3 SD of target height;
* Syndrome disorders with or without mental retardation;
* Use of anti-hyperglycaemic drugs;
* Pregnancy (pregnancy test will be performed, if applicable);
* (History of) alcohol abuse;
* Impaired renal and/or hepatic function (defined as GFR < 80 ml/min. GFR=40 x length (cm) / serumcreatinin (μmol/l and ALAT >150% of normal value for age);
* Use of ritonavir; use of ACE inhibitors;
* Insufficient knowledge of the Dutch language.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change in BMI from baseline | 18 months and 36 months
  Change in BMI after part 1 (double blind) and part 2 ( follow-up)
Change in Insulin resistance from baseline | 3; 6; 9; 12; 15; 18; 24; 30 and 36 months
  calculated by the Homeostasis Model Assessment for Insulin Resistance (HOMA-IR).

SECONDARY OUTCOMES:
Renal and hepatic function | 3; 6; 9; 12; 15; 18; 24; 30 and 36 months
  creatinine and alat
Tolerability | 3; 6; 9; 12; 15; 18; 24; 30 and 36 months
  The amount of reported adverse effects, in relation to the achieved dose level.
Pharmacokinetics (PK)-parameters: clearance (ml/min) | 9 months
  Clearance where applicable expressed per body weight, age category, Tanner Stage and gender, clearance will be determined with a two-compartment pharmacokinetic model using non linear mixed effect modelling.
Body fat percentage | 0, 9, 18 and 36 months
Physical fitness | 0, 9, 18 and 36 months
Quality of life | 0, 9, 18 and 36 months
Long term efficacy | 36 months
  Based on BMI and HOMA-IR values
Long-term safety | 36 months
  Renal and hepatic function after 36 months of metformin use
Long-term tolerability | 36 months
  The amount of adverse effects after 36 months
Microvascular complications | 36 months
  Measured as micro-albuminuria
Macrovascular complications | 36 monthts
  Measured with Pulse Wave Velocity and Augmentation Index.
Development of T2DM | 36 months
PK-parameters: volume of distribution (liters) | 9 months
  Volume of distribution, where applicable expressed per body weight, age category, Tanner Stage and gender, volume of distribution will be determined with a two-compartment pharmacokinetic model using non linear mixed effect modelling.

CONTACTS AND LOCATIONS:
Overall Officials: Marja MJ van der Vorst, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - St. Antonius Hospital, Nieuwegein

REFERENCES:
- [Derived] van Rongen A, van der Aa MP, Matic M, van Schaik RHN, Deneer VHM, van der Vorst MM, Knibbe CAJ. Increased Metformin Clearance in Overweight and Obese Adolescents: A Pharmacokinetic Substudy of a Randomized Controlled Trial. Paediatr Drugs. 2018 Aug;20(4):365-374. doi: 10.1007/s40272-018-0293-1. PMID 29748932
- [Derived] van der Aa MP, Hoving V, van de Garde EM, de Boer A, Knibbe CA, van der Vorst MM. The Effect of Eighteen-Month Metformin Treatment in Obese Adolescents: Comparison of Results Obtained in Daily Practice with Results from a Clinical Trial. J Obes. 2016;2016:7852648. doi: 10.1155/2016/7852648. Epub 2016 Dec 22. PMID 28101379
- [Derived] van der Aa MP, Elst MA, van Mil EG, Knibbe CA, van der Vorst MM. METFORMIN: an efficacy, safety and pharmacokinetic study on the short-term and long-term use in obese children and adolescents - study protocol of a randomized controlled study. Trials. 2014 Jun 5;15:207. doi: 10.1186/1745-6215-15-207. PMID 24899137